CLINICAL TRIAL: NCT07255833
Title: Retrospective Analysis of ECG Changes and Arrhythmias in Patients With Profound Hyponatremia
Status: Completed | Type: Observational
Sponsor: University of Cologne (Other)
Responsible Party: Principal Investigator, Volker Burst, Prof. Dr. med, University of Cologne
Other Study IDs: Retro-EKG
Record Dates: First submitted 2025-09-22; First posted 2025-12-01 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Hyponatremia
Keywords: hyponatremia; ECG; arrhythmias; cardiac; conduction
MeSH Terms: conditions — Hyponatremia; Arrhythmias, Cardiac

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The primary objective of this retrospective study is to determine the impact of hyponatremia on quantitative measurements and characteristics of the ECG. Secondary objectives comprise qualitative ECG features during hyponatremia, such as lead type, rhythm, etc.

DETAILED DESCRIPTION:
Hyponatremia is the most common electrolyte disorder in hospitalized patients. It is associated with high morbidity and mortality. Acute profound hyponatremia is defined by a drop in sodium level to < 125 mEq/L within ≤ 48 h. As the cation with the highest extracellular concentration, sodium is the main determinant of serum osmolality. Thus, profound hyponatremia can lead to hypoosmolality of the serum (< 275 mosmol/kg) and a resulting osmotic gradient to a variably pronounced cerebral edema with neurological and/or psychiatric symptoms such as confusion, nausea, psychosis, vigilance disorder up to coma or seizures.

While the effects of hyponatremia on the central nervous system (CNS) are well characterized, its effects on cardiac function, particularly excitation and conduction system, are poorly understood. Thus, it is unclear whether osmotically induced swelling of human cardiomyocytes is a possible pathophysiological mechanism for cardiac dysfunction. In animal studies with isolated ventricular cardiomyocytes from rabbit hearts, significant swelling of cardiomyocytes was shown under osmotic stress in both ischemic preconditioned and non-preconditioned cells. In another experimental study, Yanagi et al. systematically investigated the effects of decreasing extracellular sodium concentration on the mechanical and electrophysiological properties of pig hearts in the Langendorff perfusion model. Electrocardiographic changes in the PQ interval and QT duration were demonstrated with decreasing sodium concentration as an expression of impaired atrioventricular and intraventricular conduction.

In contrast, there are no clinical cohort studies in which the frequency and prognostic relevance of electrocardiographic changes and arrhythmias in profound hyponatremia have been investigated. The majority of publications comprise case reports and small case series describing variable and mostly reversible electrocardiographic changes and arrhythmias associated with profound hyponatremia.

The electrocardiogram (ECG) as a primary basic diagnostic tool plays a central role in cardiology and emergency medicine in particular for clarifying chest pain, shortness of breath, palpitations and dizziness/syncope. In addition, it can also provide indications of pathologies outside the cardiovascular system such as intoxication or electrolyte disorders or be used to monitor drug therapy.

The extent to which the ECG can be used in the diagnosis and risk stratification of profound hyponatremia cannot be answered today, but the aforementioned case reports suggest that hyponatremia might have an influence on the electrophysiological processes of the heart and thus the ECG.

The primary objective of this retrospective study is to determine the impact of hyponatremia on quantitative measurements and characteristics of the ECG. Secondary objectives comprise qualitative ECG features during hyponatremia, such as lead type, rhythm, etc. All ECG are evaluated by cardiologists as well as an automated AI application during and after resolution of hyponatremia.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients ≥18 years of the Emergency Department of the University Hospital of Cologne/Germany
* Plasma sodium ≤125 mmol/L in the admission blood sample and ≥ 130 mEq/L in a subsequent sample obtained during inpatient care.
* 12-lead-ECG on admission and a second ECG during inpatient care after resolution of profound hyponatremia.

Exclusion Criteria:

* Lack of follow-up sodium analyses within the first 24 hours after admission
* initial blood glucose >300 mg/dL
* Moderate or severe hypokalemia (potassium level < 3 mmol/L)
* Moderate or severe hyperkalemia (potassium level > 6 mmol/L)
* Pacemaker dependency with ventricular pacing
* Relevant structural heart disease
* Severe ischemic cardiomyopathy with an EF < 35%
* Untreated severe aortic valve stenosis
* Dilated cardiomyopathy (DCM)
* Hypertrophic cardiomyopathy (HCM)
* Arrhythmogenic right ventricular cardiomyopathy (ARVC)
* Infiltrative cardiomyopathy
* Ion channel disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with profound hyponatremia presenting to the emergency department
Sampling Method: Non-Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-01-01 (Actual)

PRIMARY OUTCOMES:
Comparison of quantitative (numeric) ECG features during and after resolution of hyponatremia. | at baseline and up to 1 year
  The primary aim is to determine the influence of hyponatremia on numeric ECG features of cardiac conduction (i.e., heart rate [beats per minute, bpm], RR interval [milliseconds, ms], PQ interval [ms], QRS duration [ms], (corrected) QT duration [ms], T-Wave [millimeters, mm], changes in ST segment, including ST elevations [mm] (STEMI mimics), ST depressions [mm]) in a large cohort of patients in the emergency department (ED). It is also to determine in a before-after comparison whether these features changed after correction of profound hyponatremia.

SECONDARY OUTCOMES:
Comparison of qualitative ECG features during and after resolution of hyponatremia. | at baseline and up to 1 year
  Secondary outcome measures comprise qualitative (non-numeric) characteristics of the ECG waveform, such as ECG lead type, rhythm, changes in ST segment, including ST elevations (STEMI mimics), ST depressions, T wave inversions, block patterns, conduction disturbances, Brugada-typical changes, etc. in the same ED cohort during hyponatremia. A before-after comparison was performed to assess whether these features changed after correction of profound hyponatremia.
Detection of hyponatremia on the basis of ECG changes. | at baseline
  To determine the sensitivity and specificity of the ECG for profound hyponatremia.

CONTACTS AND LOCATIONS:
Overall Officials: Volker Burst, MD, Prof, Principal Investigator — University Hospital Cologne
Locations (1):
- University Hospital Cologne, Cologne, Germany

IPD SHARING:
Plan to Share IPD: Yes
Data base will be shared upon request